CLINICAL TRIAL: NCT02368990
Title: T-STAR - T790M Mutation Positive 2nd Line STandard of cAre Registry
Brief Title: T790M Mutation Positive 2nd Line STandard of cAre Registry
Acronym: T-STAR
Status: Withdrawn | Type: Observational
Why Stopped: Since the conception of the study, the competitive environment has developed and as a result this study is no longer able to generate the necessary information.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160R00001
Record Dates: First submitted 2015-01-29; First posted 2015-02-23 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; T790M; EGFR; TKI Resistance; Non Small Cell Lung Cancer; AZD9291; Clovis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSCLC T790M positive: NSCLC patients who have had 1st line treatment with an approved EGFR targeted TKI, who are known to be T790M mutation positive and who have been prescribed platinum based doublet chemotherapy (pemetrexed + cisplatin/carboplatin) as a 2nd line treatment as part of their standard care.

SUMMARY:
The aim of the study is to collect real world information on patients with locally advanced or metastatic non small cell lung cancer (NSCLC) who progressed after first line treatment with an approved Tyrosine-Kinase Inhibitor (TKI), who are known to be T790M positive and have been prescribed second line platinum-based chemotherapy (Pemetrexed + Cisplatin /Carboplatin).

DETAILED DESCRIPTION:
The study is an observational prospective cohort study that plans to enroll approximately 200 patients worldwide. There are Epidermal Growth Factor Receptor (EGFR) mutations known to be associated with EGFR-targeted TKI sensitivity ( Ex19Del, L858R, L861Q, and G719X). Further tests on biopsied tissue or cytology at progression after treatment with an approved EGFR targeted TKI are used to determine positivity to T790M mutation. Primary objectives of the study are :

* To estimate overall survival
* To estimate disease progression (as assessed and defined by physician)
* To estimate time on treatment by line of therapy
* To describe time to subsequent therapies (or death)
* To describe healthcare resource utilization patterns
* To capture patient reported symptoms, functioning, and health-related quality of life (HRQoL) data using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 items (EORTC QLQ-C30) and European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 items (EORTC QLQ-LC13)
* To describe the use of pemetrexed + cisplatin/carboplatin as the 2nd line treatment
* To describe treatment patterns for 3rd line treatment and beyond

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent prior to any study specific procedure.
* Patients with histologically- or cytologically-documented NSCLC who present with Stage IIIB/ Stage IV disease.
* Evidence of radiological disease progression following 1st line treatment for advanced/metastatic NSCLC with an approved EGFR-targeted TKI monotherapy without any additional concurrent NSCLC treatment. Chemotherapy received in the adjuvant setting is permitted.
* Patients prescribed platinum based doublet chemotherapy (pemetrexed + cisplatin/carboplatin) for 2nd line treatment of NSCLC. Treatment must have been selected by physician as part of routine standard of care, prior to confirming eligibility for the study. Patient must be enrolled into the study within two cycles of beginning treatment. Treatment must be given in accordance with local prescribing information.
* Confirmation prior to enrolment into the study that the tumour harbours the following EGFR mutations known to be associated with EGFR-targeted TKI sensitivity: Ex19Del, L858R, L861Q, and G719X.
* Patients must have had confirmation that tumour is T790M mutation positive from a biopsy or cytology sample taken after confirmed disease progression on 1st line treatment with an approved EGFR-targeted TKI.
* WHO performance status 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.

Exclusion Criteria:

* Treatment with any of the following:

  * Prior treatment with more than one line of treatment for advanced NSCLC.
  * Major surgery (excluding placement of vascular access) within 4 weeks prior to enrolment.
  * Palliative radiotherapy with a limited field of radiation within 1 week prior to enrolment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks prior to enrolment.
* Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to enrolment.
* Patients who are known to be entering an alternative interventional clinical study at the time of enrolment into this study will be excluded. However, inclusion in this study does not preclude participation in any other clinical study after enrolment. Patients who participate in clinical studies after enrolment into this study will be followed to the extent possible as permitted by the sponsor of that clinical study.
* Involvement in the planning and conduct of the study (applies to AstraZeneca staff or staff at the site).
* Judgment by the physician that the patient should not participate in the study if the patient is unlikely to comply with procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed EGFRm+, T790M mutation positive, locally advanced or metastatic NSCLC who have been prescribed pemetrexed + cisplatin/carboplatin in accordance with clinical practice after 1st line treatment with approved EGFR-targeted TKI will be selected from approximately 100 sites across 17 countries worldwide.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 24 months from last subject in
  This will be assessed as the time from the start date of 2nd line chemotherapy until death due to any cause or censoring (at end of 24 months).To assess efficacy of permetrexed + cisplatinum/carboplatin as the 2nd line of treatment of NSCLC.

SECONDARY OUTCOMES:
Response to Therapy as assessed by the physician | 24 months from last subject in
  This will be assessed as the time from start of 2nd line therapy until the date of disease progression or death (by any cause in the absence of progression). To assess efficacy of 2nd line treatment and beyond.
Time on treatment by line of therapy and between therapies | 24 months from last subject in
  This will be assessed as the time from start date of line of therapy to end date of line of therapy or death date. To describe treatment patterns for 2nd line and beyond.
Admission of planned/unplanned hospitalizations, emergency department visits and outpatient/physician visits | 24 months from last subject in
  This will be assessed as the number and Time from the dates of admission and exit of attendance. To describe Healthcare resource utilization for 2nd line treatment and beyond.
Time to symptom deterioration | 24 months from last subject in
  For each of the symptoms in EORTC QLQ-LC13 and EORTC QLQ-C30, Time from inclusion until the date of first clinically meaningful symptom deterioration or death by any cause in the absence of a clinically meaningful symptom deterioration. To assess the impact of 2nd and subsequent lines of therapy on patients' disease-related symptoms and health related quality of life.
Symptom Improvement Rate | 24 months from last subject in
  This will be assessed as the number of patients with two consecutive assessments, which showed a clinically meaningful improvement in that symptom from baseline. To assess the impact of 2nd and subsequent lines of therapies on patients' disease-related symptoms and health related quality of life.
Duration of Response as defined by the physician | 24 months from last subject in
  This will be assessed as the time from the date of complete or partial response until the first date of recurrence or progression. To assess the efficacy of 2nd line treatment and beyond.
Progression Free Survival | 24 months from last subject in
  This will be assessed as the time from start of 2nd line therapy until the date of disease progression or death by any cause. This will be done to assess efficacy of pemetrexed + cisplatin/carboplatin as the 2nd line treatment of NSCLC.

CONTACTS AND LOCATIONS:
Locations (49):
- United States (3):
  - Research Site, Kentucky, Kentucky
  - Research Site, Maryland City, Maryland
  - Research Site, Langhorne, Pennsylvania
- China (9):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Jiangsu
  - Research Site, Jilin
  - Research Site, Shanghai
  - Research Site, Shanghai Ruijin Hospital
  - Research Site, Sichuan Cancer Hospital
  - Research Site, Xi'an
- France (7):
  - Research Site, Boulogne-Billancourt
  - Research Site, Bretagne
  - Research Site, La Chaussée-Saint-Victor
  - Research Site, Lille
  - Research Site, Pontoise
  - Research Site, Rhone-Alpes
  - Research Site, Saint-Quentin
- Research Site, Esslingen am Neckar, Germany
- Italy (10):
  - Research Site, Catania
  - Research Site, Ferrara
  - Research Site, Messina
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Rome
  - Research Site, Torino
- Research Site, Groningen, Netherlands
- Russia (2):
  - Research Site, Barnaul
  - Research Site, Saint Petersburg
- Spain (13):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, León
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Ourense
  - Research Site, Pamplona
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Vizcaya
- Taiwan (3):
  - Research Site, Linkou District
  - Research Site, Taichung
  - Research Site, Taipei